CLINICAL TRIAL: NCT06663124
Title: Extreme Capsule Electrical Stimulation for Drug-resistant Focal Epilepsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liankun_Ren, Professor, Xuanwu Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-083
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Epilepsy, Drug Resistant
Keywords: Extreme capsule; Deep Brain Stimulation; Drug Resistant Epilepsy; Focal Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsies, Partial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EC-DBS group (Experimental): participants will undergo EC-DBS ON with the individual stimulation parameters determined in the parameter determination period, then continue to receive stimulation for the remainder of the study.
  Interventions: Device: EC-DBS ON

INTERVENTIONS:
Device: EC-DBS ON — The surgical intervention named deep brain stimulation is a well-established neurosurgical treatment for drug-resistant epilepsy.The targets used in this study are extreme capsule.The devices used for intervention have been approved by Chinese National Medical Products Administration (CFDA). The postoperative drug dosage adjustment depends on the efficacy of DBS and the judgment of the epilepsy specialist.

SUMMARY:
Evaluation of the Efficacy and Safety of Deep Brain Stimulation of the Extreme Capsule (EC) for the Treatment of Drug-Resistant Epilepsy

DETAILED DESCRIPTION:
This studyTo evaluate the efficacy and safety of deep brain stimulation of the EC for the treatment of drug-resistant epilepsy originating from EC structurally connected cortex cortex, This study aims to explore stimulation patterns and parameters that can suppress abnormal epileptic discharges at the seizure focus without impairing language function. This study aims to improve treatment challenges for these patients and promote clinical translation and application

ELIGIBILITY:
Inclusion Criteria:

* Participants are between the ages of 14 -65 years of age
* Diagnosis of drug-resistant epilepsy follows the standard of resistance to regular medication treatment for at least two years. Comprehensive preoperative epilepsy assessment, combined with individualized fiber tracking, is used to determine whether the epileptogenic zone is located in cortex regions structurally connected to the extreme capsule.
* Persistence of disabling seizures at least 3 times per month or greater,
* Informed consent signed.

Exclusion Criteria:

* Structural alterations are present in the extreme capsule.
* Diagnosed with generalized or hereditary epilepsy with ion channel gene mutations;
* Psychogenic non-epileptic seizures within 12 months;
* Presence of implanted electrical stimulation medical device anywhere in the body (e.g., pacemaker, spinal cord stimulator, responsive neurostimulation) or any metallic implants in the head (e.g., aneurysm clips, cochlear implants). Note: Vagal nerve stimulators are allowed if the parameter remains stable for at least 3 months prior to the screening visit;
* Risk factors that would put the participant at risk for intraoperative or postoperative bleeding. (e.g., coagulation abnormalities, etc.) or the need for chronic anticoagulation or antiplatelet aggregation medications;
* IQ < 55 or severe cognitive dysfunction, unable to complete the study;
* Diagnosed with a progressive neurological disorder (including progressive Rasmussen's encephalitis, etc.);
* Diagnosed with a severe neuropsychiatric disorder such as dementia, major depression (admission to a psychiatric specialty/hospital within 5 years or any suicidal or self-injurious tendencies), schizophrenia, or neurodegenerative disorders;
* Diagnosed with other serious physical disorders, internal diseases or severe abnormalities in liver or kidney function;
* Pregnant, or planning to pregnant within 2 years;
* Participation in another clinical study within 3 months;
* Not suitable for enrollment as assessed by the multidisciplinary team of the center.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency (SF28) | Up to 1 year after EC-DBS
  Seizure frequency (SF28) is defined as seizure count per month (28-day) period. The SF28 is calculated as follows, where D=total number of days for which seizure information is collected for the specific 28-day interval:
  SF28=(Total number of seizures in D days/D)*28. In addition, the baseline seizure frequency is defined as mean of 3-month SF28 in the baseline period. The seizure frequency in double-blind phase is defined as SF28 per month during the double-blind period. Percent change in seizure frequency=100*(double-blind SF28-baseline SF28)/baseline SF28.

SECONDARY OUTCOMES:
Seizure Responder Rate | Up to 1 year after EC-DBS
  The proportion of patients with a ≥ 50% reduction from Baseline in seizure frequency.
Life quality evaluation | Up to 1 year after EC-DBS
  Percentage change from baseline in Quality of Life in Epilepsy-31 inventory (QOLIE-31) score.
Adverse Events | Up to 1 year after EC-DBS
  Rate of adverse events which were judged to be study-related throughout the study.
Incidence of Sudden Unexpected Death in Epilepsy (SUDEP) | Up to 1 year after EC-DBS
  The number presented is for Definite and Probable SUDEP. The rate is calculated per 1000 subject years of follow

CONTACTS AND LOCATIONS:
Overall Officials: Liankun Ren, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No